CLINICAL TRIAL: NCT00374413
Title: Clinical Study Protocol for the Investigation of the Kineflex|C Spinal System - a Pivotal Study in Continued Access Stage
Brief Title: Kineflex|C Artificial Disc System to Treat Cervical Degenerative Disc Disease (DDD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Economic and business factors
Sponsor: SpinalMotion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kineflex|C
Record Dates: First submitted 2006-09-07; First posted 2006-09-11 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-08

CONDITIONS: Degenerative Disc Disease (DDD)
Keywords: DDD; artificial disc
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Total Disc Replacement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kineflex-C (Experimental)
  Interventions: Device: Artificial disk; Device: Artificial disc
- ACDF (Active Comparator)
  Interventions: Device: Artificial disk; Device: Artificial disc

INTERVENTIONS:
Device: Artificial disk — Implant
Device: Artificial disc — Implant

SUMMARY:
The purpose of this study is to show that the Kineflex|C Spinal System is no worse than conventional Anterior Cervical Diskectomy with Fusion (ACDF) in patients with single level degenerative disc disease at any cervical level from C3 to C7.

DETAILED DESCRIPTION:
The Kineflex|C disc is a 3-piece modular design consisting of two cobalt chrome molybdenum (CCM) end-plates and a fully articulating CCM core. The system is available in two foot print sizes.

ELIGIBILITY:
Inclusion Criteria:

* have symptoms of cervical degenerative disc disease (DDD) at only one cervical level from C3 to C7, disc herniation on CT or MRI;
* have radiculopathy symptoms in neck, one or both shoulders, and/or one or both arms;
* have at least six months of prior conservative treatment (e.g., physical therapy and/or use of anti-inflammatory medications and muscle relaxants at the manufacturer's recommended therapeutic dose), the presence of progressive symptoms (e.g., increasing numbness or tingling), or signs of nerve root compression;
* have moderate disability neck disability index (NDI) score; AND
* be likely to return for all follow-up visits and be willing and able to provide informed consent for study participation

Exclusion Criteria:

* marked cervical instability;
* non discogenic neck pain or non discogenic source of symptoms;
* radiographic confirmation of severe facet disease or facet degeneration;
* bridging osteophytes;
* prior surgery at the level to be treated;
* prior fusion at any cervical level;
* more than one neck surgery via anterior approach;
* previous trauma to the C3-C7 levels resulting in compression or bursting;
* documented presence of free nuclear fragment at any cervical level;
* severe myelopathy;
* any paralysis;
* history of chemical or alcohol dependence;
* active systemic infection;
* infection at the site of surgery;
* prior disc space infection or osteomyelitis in the cervical spine;
* any terminal, systemic or autoimmune disease;
* metabolic bone disease (e.g., osteoporosis, gout, osteomalacia, Paget's disease);
* any disease, condition or surgery which might impair healing;
* known metal allergy;
* arachnoiditis;
* currently experiencing an episode of major mental illness;
* pregnancy at time of enrollment, or planning to become pregnant, since this would contraindicate surgery;
* morbid obesity; use of spinal stimulator at any cervical level prior to surgery;
* currently a prisoner;
* currently involved in spinal litigation which may influence the subjects reporting of symptoms; OR
* lives more than 300 miles from study center or participation in any other investigational drug, biologic, or medical device study within the last 30 days prior to study surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 343 (Actual)
Dates: Start 2005-07; Primary Completion 2010-01 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Improvement in Neck Disability Index (NDI) Score at 24 months compared with baseline | 24 months
No major device related adverse events | 24 months

SECONDARY OUTCOMES:
Clinically significant improvement in one or more radicular symptoms at 24 months compared to baseline | 24 months
Time to recovery | 24 months
Disc height at 24 months compared to baseline | 24 months
Adjacent level deterioration at 24 months compared to baseline | 24 months
Progressive facet disease at 24 months compared to baseline | 24months
Displacement or migration of the device | 24 months
Odom's Criteria | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Fred Geisler, MD, Principal Investigator — Medical Monitor
Locations (21):
- United States (21):
  - Tower Orthopedics and Sports Medicine, Beverly Hills, California
  - Kaiser Foundation Research Institute, Oakland, California
  - University of California San Diego, San Diego, California
  - Rocky Mountain Associates in Orthopedic Medicine, P.C., Loveland, Colorado
  - Emory Orthopaedics & Spine Center, Atlanta, Georgia
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - Maryland Brain and Spine Center, Annapolis, Maryland
  - Orthopaedic Associates, P.A, Towson, Maryland
  - William Beaumont Hospital, Royal Oak, Michigan
  - Sierra Regional Spine Institute, Reno, Nevada
  - Hamilton Orthopaedic Surgery and Sports Medicine, Hamilton, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Manhattan Orthopaedics, P.C., New York, New York
  - Carolina Neurosurgery and Spine Associates, Charlotte, North Carolina
  - Triangle Orthopaedic Associates, P.A., Durham, North Carolina
  - Univ. of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Semmes-Murphy Clinic, Memphis, Tennessee
  - Plano Orthopedic Sports Medicine & Spine Center, Plano, Texas
  - SpineMark CRO at Texas Back Institue, Plano, Texas
  - Gordon Spine Associates, Tyler, Texas
  - Orthopedics International Spine, Kirkland, Washington

REFERENCES:
- [Derived] Coric D, Guyer RD, Nunley PD, Musante D, Carmody C, Gordon C, Lauryssen C, Boltes MO, Ohnmeiss DD. Prospective, randomized multicenter study of cervical arthroplasty versus anterior cervical discectomy and fusion: 5-year results with a metal-on-metal artificial disc. J Neurosurg Spine. 2018 Mar;28(3):252-261. doi: 10.3171/2017.5.SPINE16824. Epub 2018 Jan 5. PMID 29303467
- [Derived] Coric D, Nunley PD, Guyer RD, Musante D, Carmody CN, Gordon CR, Lauryssen C, Ohnmeiss DD, Boltes MO. Prospective, randomized, multicenter study of cervical arthroplasty: 269 patients from the Kineflex|C artificial disc investigational device exemption study with a minimum 2-year follow-up: clinical article. J Neurosurg Spine. 2011 Oct;15(4):348-58. doi: 10.3171/2011.5.SPINE10769. Epub 2011 Jun 24. PMID 21699471
- See also: Related Info — http://www.spinalmotion.com